CLINICAL TRIAL: NCT05334485
Title: Pyridostigmine Efficacy and Safety for Treatment of Ileus After Colorectal Surgery (PESTI Trial)
Brief Title: Pyridostigmine Efficacy and Safety for Treatment of Ileus After Colorectal Surgery
Acronym: PESTI
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stefan Holubar MD MS FACS, FASCRS (Other)
Responsible Party: Sponsor-Investigator, Stefan Holubar MD MS FACS, FASCRS, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-915
Record Dates: First submitted 2022-03-09; First posted 2022-04-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — Pyridostigmine Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pyridostigmine (Experimental): Patients randomized to this group will be given 60mg of pyridostigmine bromide orally, every 12 hours. Pyridostigmine will be administered from the time of diagnosis of postoperative ileus until the return of bowel function, or for a maximum of 48 hours.
  Interventions: Drug: Pyridostigmine Bromide
- Placebo (Placebo Comparator): Patients randomized to this group will be given starch orally, every 12 hours for a maximum of 48 hours.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pyridostigmine Bromide — Oral 60mg pyridostigmine bromide
  Arms: Pyridostigmine
Other: Placebo — Oral starch placebo
  Arms: Placebo

SUMMARY:
A double blind, placebo controlled, randomized control trial studying the safety and efficacy of pyridostigmine as a rescue therapy for postoperative ileus. Patients who undergo elective colorectal resection with or without creation of an ostomy, and subsequently develop postoperative ileus will be eligible for enrollment. Patients will be randomized to receive either pyridostigmine or placebo in addition to the current elements of standard of care. Patients will also complete the pyridostigmine bromide side effects scale (PBSES) upon enrollment and following each administration of either intervention or placebo to monitor treatment safety and evaluate for the development of side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age 18 and over) patients with benign or malignant colonic or rectal disease who have undergone elective laparoscopic, robotic, or open colorectal resections with or without ostomy construction at our center, and subsequently developed POI, defined as symptoms of bloating with or without nausea and vomiting, with absence of passage of flatus or stool for at least 48 hours postoperatively and require return to NPO status after initial diet attempts with or without placement of an NGT.
2. Radiographic confirmation of POI diagnosis either via abdominal radiography (KUB), computed tomography abdomen/pelvis (CT A/P), or both
3. ECOG Performance status < 4
4. Laboratory evidence of normal organ function, defined as:

   1. Hemoglobin ≥ 7.0 g/dL
   2. WBC ≤ 20,000/mcL and ≥ 4,000/mcL
   3. Platelet count ≥ 100,000/mcL or ≤ 100,000,000/mcL
   4. AST (SGOT) ≤ 2.5 times the institutional upper limit of normal
   5. ALT (SGPT) ≤ 2.5 times the institutional upper limit of normal
   6. Total bilirubin within the upper limit of institutional normal range
   7. Serum Creatinine within the upper limit of institutional normal range

Exclusion Criteria:

1. Radiographic evidence of bowel obstruction
2. Documented intraabdominal septic complications (IASC, such as abdominopelvic abscess, peritonitis, anastomotic leak) at any time prior to or after enrollment
3. Isolated small bowel or ostomy surgery without colon or rectal resection
4. ASA score 5
5. Pregnant or breastfeeding females as PYR is classified by the FDA as a pregnancy risk category C medication with the potential for teratogenic or abortifacient effects and demonstrated secretion into breastmilk with an unknown but potential risk for adverse effects in the nursing infants
6. Current use of any other investigational agents including: neostigmine or other acetylcholine esterase inhibitors, alvimopan, metoclopramide, erythromycin, methylnaltrexone, naloxegol, cisapride, and laxatives or cathartics (i.e. milk of magnesia, polyethylene glycol)
7. History of allergic reactions attributed to PYR or other acetylcholine esterase inhibitors
8. Patients with any of the following uncontrolled, concurrent illnesses: active or latent MG, bronco-constrictive disease (asthma/reactive airway disease), chronic obstructive lung disease (COPD), symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia including bradycardia, renal failure, hepatic failure, gastroparesis, short bowel syndrome (small bowel < 200cm), preexisting short or large bowel dysmotility or pseudo-obstruction, chronic constipation/laxative use, peritoneal carcinomatosis, and psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Time until return of bowel function | Time from administration of pyridostigmine bromide or placebo until first passage of flatus for up to 30 days
  Following the administration of either pyridostigmine bromide or placebo, the time (in minutes) until return of bowel function will be recorded. Return of bowel function is defined as the first passage of flatus.
Incidence of pyridostigmine bromide associated side effects | Participants will complete the survey at enrollment and then again at 30 minutes following each administration of either pyridostigmine bromide or placebo.
  Side effects of pyridostigmine bromide will be assessed using the Pyridostigmine Bromide Side Effects Scale (PBSES) survey tool. Participants will complete this survey at specific time points to evaluate and monitor for the development of established side effects associated with pyridostigmine bromide administration.

SECONDARY OUTCOMES:
Time to passage of stool after postoperative ileus diagnosis | Time from the point of postoperative ileus diagnosis until the first passage of stool for up to 30 days
  The amount of time (in minutes) from the participant being diagnosed with postoperative ileus confirmed with imaging findings until the first passage of stool.
Time to tolerance of solid food after postoperative ileus | Time from the point of postoperative ileus diagnosis until first meal in which solid food is tolerated for up to 30 days
  The amount of time (in minutes) from the participant being diagnosed with postoperative ileus confirmed with imaging findings until the first tolerance of solid food.
Number of participants with complications | 30-day period following surgery
  The number of participants with any type of complication or adverse event occurring within the first 30-days following surgery.
Number of participants requiring re-operation | 30-day period following initial surgery
  The number of participants who require a re-operation for any reason during the first 30-days following the initial operation.
Number of participants requiring re-admission | 30-day period following surgery
  The number of participants requiring re-admission to the hospital for any reason during the first 30-days following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan D Holubar, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No